CLINICAL TRIAL: NCT02734043
Title: Roadmap for Succeeding in Bundled Payment for Orthopedic Joint Replacements
Status: Withdrawn | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Amol Navathe, MD, PHD, University of Pennsylvania
Other Study IDs: 824614
Record Dates: First submitted 2016-03-31; First posted 2016-04-12 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Osteoarthritis
Keywords: bundled payment
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the study is to provide a road map that can help organizational leaders understand how to sequence their financial and human capital investments related to bundled payment arrangements. Although specific strategies will vary between organizations, providing evidence from a health system with extension experience bundling care for orthopedic joint replacements can be instructive for other providers entering new building arrangements. Insights from the experience of the health system can help other organizations prioritize effort and focus energy around strategies that increase the likelihood of succeeding under Comprehensive Care for Joint Replacement (CJR) and other bundled payment contracts.

DETAILED DESCRIPTION:
This study will analyze data from a health system with the longest standing experience with bundled payments for orthopedic procedures. The goal of this work is to provide insights from this health system's six years of experience and offer a road map that other organizations around the country can use as they plan and implement their own bundled payment programs. The investigators will conduct a retrospective analysis on quality and cost data from a health system with extensive experience with bundled payments for orthopedic joint replacements. The study design will consist of three parts: first, the team will report trends in quality and cost outcomes over time using descriptive statistics; second, the team will perform multi-variable regression analyses on the data to identify significant predictors of different quality and cost outcomes and provide statistical tests on the trends; third, the team will evaluate changes in physician and hospital level variation along the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* participants in this study will be physicians participating in the bundled payment arrangement at the health system in question. All physicians will be included in the analysis.

Exclusion Criteria:

* no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Orthopedic surgeons from one health system who participated over a five year span in bundled payment arrangements
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Surgical site infection at the physician level | 12 months
  The study team will evaluate at the physician level. The quality metric evaluated will be average rate of surgical site infections.

SECONDARY OUTCOMES:
Cost of care during hospitalization | 12 months
  The study team will measure secondary cost outcome variables on the episode level. The cost metric to be evaluated is per episode costs of care during the hospitalization in which the surgery occurred.
Cost of care post-discharge | 12 months
  The study team will measure secondary cost outcome variables on the episode level. The cost metric to be evaluated is per episode costs of care post-discharge.
All-cause readmission rate at the physician level | 12 months
  The study team will evaluate at the physician level. The quality metric measured will be all-cause readmission rate.
Venous thromboembolism at the physician level | 12 months
  The study team will evaluate at the physician level. The quality metric measured will be the rate of venous thromboembolism per physician in each quarter of analysis.
Cost of care at the physician level | 12 months
  The study team will evaluate at the physician level. The cost metric evaluated will be the average costs of care during hospitalization in which the surgery occurred.
Spending at the physician level | 12 months
  The study team will evaluate at the physician level. The cost metric evaluated will be average spending on care in combined hospitalization and post-discharge periods per physician in each quarter of analysis.

IPD SHARING:
Plan to Share IPD: No